CLINICAL TRIAL: NCT02212925
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses (0.5, 2.5, 10 and 20 mg q.d. for 10 Days) of BI 14332 CL as Tablet in Female and Male Patients With Type 2 Diabetes (Randomised, Double-blind, Placebo-controlled Within the Dose Groups), Followed by a 4-week Treatment Part* (Randomised, Double-blind, Placebo-controlled) of Two Doses (Planned 5 and 20 mg) Selected on the Basis of Tolerability and DPP-4 Inhibition in the Multiple Rising Dose Part
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 14332 CL as Tablet in Female and Male Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1233.2
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- BI 14332 CL (Experimental)
  Interventions: Drug: BI 14332 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 14332 CL
  Arms: BI 14332 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 14332 CL following administration of multiple rising oral doses over 10 days in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal or hysterectomised female patients with proven diagnosis of type 2 diabetes mellitus treated with diet and exercise only, or with one oral hypoglycaemic agent besides glitazones and who are not taking the maximum approved dose
* Glycosylated haemoglobin A1 (HbA1c) ≥ 6.5% and ≤ 8.5 % at screening for patients treated with diet and exercise and/or one oral hypoglycaemic agent
* Age ≥21 and Age ≤70 years (female hysterectomised and male patients) Age ≥60 and Age ≤70 years (female postmenopausal patients)
* Body Mass Index (BMI) ≥18.5 and BMI ≤35 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including BP, pulse rate (PR) and ECG) deviating from normal and of not acceptable clinical relevance
* Clinically relevant concomitant diseases like renal insufficiency, cardiac insufficiency New York Heart Association (NYHA) II-IV, myocardial infarction, other known cardiovascular diseases including hypertension > 140/90 mmHg, stroke and transient ischemic attack
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders besides type 2 diabetes, hyperlipidaemia and medically treated hypertension
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or relevant neurological disorders besides polyneuropathy
* Chronic or relevant acute infections (e.g. HIV, Hepatitis)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial except allowed co-medication
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Antidiabetic treatment with more than one oral hypoglycaemic agent or insulin or glitazones and anti-hypertensive treatment with verapamil or diltiazem
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 40 g/day = 5 units/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Any laboratory value outside the reference range and the clinical relevance is not acceptable (or the value is more than three times higher than the upper limit of the normal range e.g. liver enzymes)
* Change of drug dosing of allowed co-medication (anti-hypertensive agents, acetylic salicylic acid and statins) within the last 3 months
* Fasted blood glucose > 240 mg/dl (>13.3 mmol/L) on two consecutive days during washout
* Serum creatinine above upper limit of normal at screening
* Male patients not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until one month after the last intake
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female patients:

* Child bearing potential
* Positive pregnancy test
* Lactation period

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 14 days after last drug administration
Number of patients with clinically significant findings in vital signs (blood pressure, pulse rate) | up to 14 days after last drug administration
Number of patients with clinically significant findings in ECG | up to 14 days after last drug administration
Number of patients with clinically significant findings in laboratory tests | up to 14 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 14 days after last drug administration

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 18 days after first drug administration
tmax (time from dosing to maximum concentration) | up to 18 days after first drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point within the first dosing interval) | up to 18 days after first drug administration
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 h after administration of the first dose) | up to 18 days after first drug administration
Ae0-24 (amount of analyte that is eliminated in urine from the time interval 0 h to 24 h) | up to 11 days after first drug administration
fe0-24 (fraction of analyte excreted in urine from time point 0 h to 24 h) | up to 11 days after first drug administration
CLR,0-24 (renal clearance of the analyte in plasma from the time point 0 h until the time point 24 h) | up to 11 days after first drug administration
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval) | up to 18 days after first drug administration
Cpre,N (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose N) | up to 18 days after first drug administration
PTF (peak trough fluctuation) | up to 18 days after first drug administration
  in percent
RA,Cmax (accumulation ratio based on Cmax) | up to 18 days after first drug administration
RA,AUC(accumulation ratio based on AUCτ) | up to 18 days after first drug administration
Change in dipeptidyl-peptidase 4 (DPP-IV) activity | baseline, up to 18 days after first drug administration
Area under the curve of plasma glucose | baseline, up to 3 hours after intake of standardized meal